CLINICAL TRIAL: NCT01898806
Title: A Phase 4 Multicenter, Randomized, Placebo Controlled Trial of 3 Doses of Intralesional Triamcinolone (KENALOG®) In the Treatment of Mild to Moderate Patch Type Alopecia Areata
Brief Title: Intralesional Steroids in the Treatment of Alopecia Areata
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The PI left the Columbia University Medical Center. Study was not Completed.
Sponsor: Columbia University (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAI5852
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Kenalog; Triamcinolone
MeSH Terms: conditions — Alopecia Areata | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- IL TAC 2.5 mg/ml (Experimental): Intralesional Triamcinolone 2.5 mg/ml (IL TAC 2.5 mg/ml):
  Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss up to the maximum dose of 30 mg IL TAC per month, for a total of 6 months. Injections will be performed at baseline, weeks 4, 8, 12, 16 and 20
  Interventions: Drug: Intralesional Triamcinolone 2.5 mg/ml
- IL TAC 5 mg/ml (Experimental): Intralesional Triamcinolone 5mg/ml (IL TAC 5 mg/ml):
  Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss up to the maximum dose of 30 mg IL TAC per month, for a total of 6 months. Injections will be performed at baseline, weeks 4, 8, 12, 16 and 20.
  Interventions: Drug: Intralesional Triamcinolone 5 mg/ml
- IL TAC 10 mg/ml (Experimental): Intralesional Triamcinolone 10mg/ml (IL TAC 10 mg/ml):
  Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss up to the maximum dose of 30 mg IL TAC per month, for a total of 6 months. Injections will be performed at baseline, weeks 4, 8, 12, 16 and 20.
  Interventions: Drug: Intralesional Triamcinolone 10 mg/ml
- Placebo (Placebo Comparator): Intralesional Saline (Placebo):
  Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss for a total of 6 months. Injections will be performed at baseline, weeks 4, 8, 12, 16 and 20. Open label treatment with IL kenalog at the dose deemed most appropriate may be administered after the 1st 6 months in nonresponders or partial responders.
  Interventions: Drug: Intralesional Saline

INTERVENTIONS:
Drug: Intralesional Triamcinolone 2.5 mg/ml — Intralesional Triamcinolone at a strength of 2.5 mg/ml. Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss up to the maximum dose of 30 mg IL TAC per month, for a total of 6 months.
  Other Names: Kenalog; IL TAC 2.5 mg/ml
  Arms: IL TAC 2.5 mg/ml
Drug: Intralesional Triamcinolone 5 mg/ml — Intralesional Triamcinolone at a strength of 5 mg/ml. Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss up to the maximum dose of 30 mg IL TAC per month, for a total of 6 months.
  Other Names: Kenalog; IL TAC 5 mg/ml
  Arms: IL TAC 5 mg/ml
Drug: Intralesional Triamcinolone 10 mg/ml — Intralesional Triamcinolone at a strength of 10 mg/ml. Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss up to the maximum dose of 30 mg IL TAC per month, for a total of 6 months.
  Other Names: Kenalog; IL TAC 10 mg/ml
  Arms: IL TAC 10 mg/ml
Drug: Intralesional Saline — Intralesional Saline (Placebo). Patients will receive intradermal injection of study medication once per month to all, or as many as possible, areas of hair loss for a total of 6 months.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study aims to determine the frequency of response to treatment with 3 concentrations of IL TAC, 2.5mg/ml, 5mg/ml or 10mg/ml as well as the duration of response and incidence of side effects compared to treatment with placebo (sterile saline solution). After the 1st 6 months, nonresponders or partial responders may be treated for 6 months with open label triamcinolone at the dose deemed appropriate by the investigator.

The investigators will also perform skin biopsies of the scalp and draw blood at selected time points in order to examine the immunohistochemical/pathological response in scalp hair follicles and the systemic circulation to treatment with IL TAC for alopecia areata.

DETAILED DESCRIPTION:
Alopecia areata (AA) is a major medical problem and is the most prevalent autoimmune disease in the US. AA represents the second most common form of hair loss and causes significant disfigurement and psychological distress to affected individuals. AA affects more individuals than most other autoimmune diseases combined, including lupus erythematosus, type 1 diabetes, psoriasis, multiple sclerosis and rheumatoid arthritis. In contrast to these conditions, research into the pathogenesis and the development of innovative therapies in AA has lagged behind.

Alopecia areata is a common form of hair loss which reportedly occurs in up to 1.7% of the population at some time in their life. Alopecia areata is apparently triggered when the individual's own immune system attacks hair follicles on the scalp or body resulting in hair loss ranging from single patches on the scalp (patch type alopecia areata) to loss of every hair on the scalp and body (alopecia universalis). Currently, there are limited treatment options for alopecia areata and unfortunately, the treatments utilized have never been rigorously tested in a placebo controlled trial.

Triamcinolone (Kenalog) is a steroid solution that has been used as a treatment for alopecia areata for over 50 years. It is administered via injection into the scalp and appears to have some efficacy for patients with mild to moderate alopecia areata. The investigators currently do not have objective data on the frequency of occurrence of successful regrowth, the duration of response or the incidence of side effects. Intralesional triamcinolone (IL TAC) is arguably the most commonly used treatments for AA, especially in patients with less than 50% hair loss. Despite this, there are no adequately powered, randomized controlled clinical trials (RCTs) examining the efficacy, safety, and duration of effect of IL TAC. In addition, the dosage or strength used varies among practitioners and the efficacy and safety of alternate doses of IL TAC has never been examined in a well designed RCT. Quantitative biomarkers for AA are a crucial step toward translational research aimed at clinical trials in AA.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 75 years of age
* Patients with a diagnosis of patch type alopecia areata
* Patients will have up to 50% total scalp hair loss at baseline as measured by the Severity of Alopecia Tool (SALT) score
* Duration of hair loss ranging from 3 to 12 months with no evidence of regrowth present at baseline in the areas to be injected

Exclusion Criteria:

* Patients with a history of or existing skin diseases affecting the scalp such as psoriasis or seborrheic dermatitis and patients with evidence of infection or skin cancer in the treated areas
* Patients in whom the diagnosis of alopecia areata is questionable
* Patients in whom regrowth is present/evident at baseline in the areas to be treated
* Patients with active medical conditions or malignancies (except adequately treated basal or squamous cell carcinoma of the skin) which in the opinion of the investigator would increase the risks associated with study participation, including patients with a history of recurrent infections
* Women of childbearing potential who are unable or unwilling to use two forms of birth control for the study duration or women who are pregnant or nursing
* Patients known to be HIV or hepatitis B or C positive or otherwise immunocompromised
* Patients with evidence of adrenal cortex abnormality or previous significant adverse reaction to intralesional steroids
* Patients unwilling or unable to discontinue treatments known to affect hair regrowth in alopecia areata
* Patients who have been treated with intralesional steroids, systemic steroids, anthralin, squaric acid, diphenylcyclopropenone (DPCP), protopic, minoxidil or other medication which in the opinion of the investigator may affect hair regrowth, within one month of the baseline visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay-Wiggan, MD, MS, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Medical Center, Department of Dermatology, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Since the PI left the institution, the only data available at this time is information on the population enrolled that was provided to the IRB. Data was not provided to the IRB per arm, but rather, for as a collective whole
Groups:
- All Participants: Includes individuals receiving intralesional triamcinolone 2.5, 5 or 10 mg/ml or intralesional placebo.
Period: Overall Study
Arm/Group | All Participants
Started | 11
Completed | 8
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Includes individuals receiving intralesional triamcinolone 2.5, 5 or 10 mg/ml or intralesional placebo. Since the PI left the institution, the only data available at this time is information on the population enrolled that was provided to the IRB. Data was not provided to the IRB per arm, but rather, for as a collective whole.
Arm/Group | All Participants
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders
Description: Comparison of the proportion of responders in each group, with response defined as 50% change (% change NOT absolute change) in SALT score from baseline (50% regrowth at week 24).
Time Frame: Up to 48 weeks
Population: Data was not collected for this outcome since enrollment was incomplete and therefore could not be analyzed. The only information available is demographics data that was submitted to the IRB for the whole group, and not stratified per arm.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Adverse Events
Description: Incidence and severity of adverse events (AEs) including the presence and degree of skin atrophy, as well as incidence of treatment-emergent laboratory abnormalities.
Time Frame: 48 weeks
Measure: Number; unit: adverse events
Arm/Group | All Participants
Number analyzed (Participants) | 8
adverse events | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- All Participants: Includes individuals receiving intralesional triamcinolone 2.5, 5 or 10 mg/ml or intralesional placebo. Data was not collected per arm, but rather, for as a collective whole.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT01898806/Prot_SAP_000.pdf